CLINICAL TRIAL: NCT03175835
Title: An Open-label, Multiple Dose, Fixed-sequence, 3-period Study to Evaluate the Drug Interaction Between CKD-519 and Rosuvastatin in Healthy Male Subjects
Brief Title: Study to Evaluate the Drug Interaction Between CKD-519 and Rosuvastatin in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 148DDI16023
Record Dates: First submitted 2017-05-18; First posted 2017-06-05 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-04

CONDITIONS: Dyslipidemias
Keywords: Dyslipidemia; CKD-519; Rosuvastatin; Drug-Drug Interaction
MeSH Terms: conditions — Dyslipidemias | interventions — Rosuvastatin Calcium; CKD-519

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rosuvastatin 20 mg & CKD-519 200 mg (Experimental): Period 1: Treatment A(Rosuvastatin 20 mg(20 mg X 1 tablet))
  Period 2: Treatment B(CKD-519 200 mg(100 mg X 2 tablets))
  Period 3: Treatment C(Rosuvastatin 20 mg(20 mg X 1 tablet), CKD-519 200 mg(100 mg X 2 tablets))
  Interventions: Drug: Rosuvastatin 20 mg; Drug: CKD-519 200 mg; Drug: Rosuvastatin 20 mg & CKD-519 200 mg

INTERVENTIONS:
Drug: Rosuvastatin 20 mg — Treatment A: Rosuvastatin 20 mg(20 mg X 1 tablet) for Day1~Day5
  Other Names: Rosuvastatin 20 mg(20 mg X 1 tablet)
Drug: CKD-519 200 mg — Treatment B: CKD-519 200 mg(100 mg X 2 tablets) for Day9~Day21
  Other Names: CKD-519 200 mg(100 mg X 2 tablets)
Drug: Rosuvastatin 20 mg & CKD-519 200 mg — Treatment C: Rosuvastatin 20 mg(20 mg X 1 tablet), CKD-519 200 mg(100 mg X 2 tablets) for Day22~Day26
  Other Names: Rosuvastatin 20 mg(20 mgX1 tablet), CKD-519 200 mg(100 mgX2 tablets)

SUMMARY:
The purpose of this study is to evaluate the drug interaction between CKD-519 and rosuvastatin in healthy male subjects.

DETAILED DESCRIPTION:
An open-label, multiple dose, fixed-sequence, 3-period study to evaluate the drug interaction between CKD-519 and rosuvastatin in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers aged between ≥ 20 and ≤ 45 years old
2. Weight ≥ 50kg, with calculated body mass index(BMI) of ≥ 18 and ≤ 29.9kg/m²
3. Subjects to consents to use effective birth controls for at least 2 months following the last dose
4. Subject is informed of the investigational nature of this study and voluntarily agrees to participate in this study and comply with the relevant instructions in written

Exclusion Criteria:

1. History or presence of clinically significant and active cardiovascular, respiratory, hepatobiliary, renal, endocrine, hematological, gastrointestinal, neurologic, immune, dermatologic or psychiatric disorder
2. With symptoms indicating acute illness within 28 days prior to the first Investigational Product administration
3. Any medical history that may affect drug absorption, distribution, metabolism and excretion
4. Any hypersensitivity reaction or clinically significant hypersensitivity reaction in the history of statin-related medication or Cholesteryl Ester Transfer Protein(CETP) inhibitor or other drugs(aspirin, antibiotics)
5. Continuous cryptogenic elevation of serum transaminase or active liver disease including elevation of serum transaminase > 3 fold upper normal limit(UNL)
6. Severe renal failure(creatinin clearance < 30 ml/min)
7. Hypothyroidism or clinically significant test result
8. Galactose intolerance, Lapp lactose intolerance, glucose-galactose malabsorption or genetic disorders
9. Any clinically significant chronic medical illness
10. Any clinically significant hypotension or hypertension (systolic < 100 mmHg/diastolic < 60 mmHg or systolic > 140 mmHg /diastolic > 90 mmHg)
11. Corrected QT interval(QTc) >450msec on 12-lead ECG
12. Positive blood tests for hemoglobins(HBs) Ag, anti-hepatitis C virus(HCV) Ab, anti-HIV Ab, or venereal disease research laboratory(VDRL)
13. Creatine phosphokinase(CPK) ≥ 5 fold of upper normal limit(UNL)
14. Use of any prescription drugs within 14 days prior to study drug administration
15. Use of any other drugs, including over-the-counter medications and herbal preparations within 7 days prior to study drug administration
16. History of clinically significant allergic reaction (However, mild allergic rhinitis or allergic dermatitis which do not require any treatment may be allowed)
17. Inability to take normal hospital diet
18. Donation of blood within 60 days prior to study drug administration or plasma to a blood bank within 20 days prior to study drug administration
19. Blood transfusion within 30 days prior to study drug administration
20. Exposure to any investigational drug or placebo within 90 days prior to the first Investigational Product(IP) administration
21. Subjects taking any drugs to induce or inhibit drug metabolizing enzymes including barbiturates within 30 days prior to the first Investigational Product(IP) administration
22. Subjects with excessive caffeine intake (more than 5 cups/day), heavy smoking (more than 10 cigarettes/day), regular alcohol intake (more than 210 g/week)
23. Subjects having been deemed inappropriate for the trial as determined by the investigator

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-06-19 (Actual); Study Completion 2017-06-19 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (Area under the plasma concentration versus time curve (AUCτ)) | 0(predose)~24 hours at Day1, Day3, Day4, Day5, Day9, Day12, Day15, Day17, Day18, Day19, Day22, Day24, Day25, Day26
  At steady state after multiple administration of CKD-519, Rosuvastatin

SECONDARY OUTCOMES:
Pharmacokinetics (Peak plasma Concentration (Cmax,ss)) | 0(predose)~24 hours at Day1, Day3, Day4, Day5, Day9, Day12, Day15, Day17, Day18, Day19, Day22, Day24, Day25, Day26
  At steady state after multiple administration of CKD-519, Rosuvastatin
Pharmacokinetics (Minimum plasma Concentration (Cmin,ss)) | 0(predose)~24 hours at Day1, Day3, Day4, Day5, Day9, Day12, Day15, Day17, Day18, Day19, Day22, Day24, Day25, Day26
  At steady state after multiple administration of CKD-519, Rosuvastatin
Pharmacokinetics (Time to maximum plasma concentration (Tmax,ss)) | 0(predose)~24 hours at Day1, Day3, Day4, Day5, Day9, Day12, Day15, Day17, Day18, Day19, Day22, Day24, Day25, Day26
  At steady state after multiple administration of CKD-519, Rosuvastatin
Pharmacokinetics (t1/2) | 0(predose)~24 hours at Day1, Day3, Day4, Day5, Day9, Day12, Day15, Day17, Day18, Day19, Day22, Day24, Day25, Day26
  At steady state after multiple administration of CKD-519, Rosuvastatin
Pharmacodynamics (CETP activity) | 0(predose)~24 hours at Day9, Day12, Day15, Day17, Day18, Day19, Day22, Day24, Day25, Day26
  At steady state after multiple administration of CKD-519, Rosuvastatin
Pharmacodynamics (CETP Concentration) | 0(predose)~24 hours at Day9, Day19, Day22, Day26
  At steady state after multiple administration of CKD-519, Rosuvastatin
Pharmacodynamics (Lipid profiles) | simultaneous with laboratory test at Day1, Day6, Day9, Day20, Day22, Day27

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No